CLINICAL TRIAL: NCT02883725
Title: National Register of Oesophageal Atresia
Acronym: REGATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: Reg 2008; 908362 (Other: CNIL number); 08.297 (Other: CCTIRS number)
Record Dates: First submitted 2016-08-18; First posted 2016-08-30 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Atresia
Keywords: Esophageal atresia
MeSH Terms: conditions — Esophageal Atresia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Esophageal atresia
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection

SUMMARY:
The esophageal atresia is a group of birth defects including a break in continuity of the esophagus with or without persistent communication with the trachea (tracheoesophageal fistula), sometimes associated (from 50%) of other malformations (heart, kidney, digestive ...).

The current prognosis for this ailment is good. However he persists a mortality (<10%) and significant morbidity, firstly related malformations (heart, kidney, for example), and secondly with particularly difficult anatomical forms (Forms long defect) .

The prevalence of this condition is estimated to be 1/2500 in 3000 live births, making an estimated ± 2,500 new cases over to 10 years in France.

The current project aims to set up a national registry (Metropolitan France and Dom Tom) to measure the prevalence of esophageal atresia among live births, phenotypic characteristics, the circumstances of their diagnosis, and their initial future at short-term during the first year of life, at which time occurs the vast majority of deaths and complications in this disease.

ELIGIBILITY:
Inclusion Criteria:

* To be born in France
* To have a esophageal atresia

Exclusion Criteria:

* To be born abroad

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All living newborns having a esophageal atresia supported in a neonatal unit, neonatal intensive care and pediatric surgery of France
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of esophageal atresia | 10 years

SECONDARY OUTCOMES:
Data collection patient with esophageal atresia | 10 years
  Circumstances of diagnosis, modalities of follow-up and clinical management
Total number of patients with complications | 10 years
Death | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Gottrand, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (37):
- France (35):
  - CHU Félix-Guyon, Saint-Denis, La Réunion
  - CHU Amiens-Picardie, Amiens
  - CHU d'Angers, Angers
  - CHRU Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - HFME de Lyon, Bron
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - CHI Créteil, Créteil
  - CHU Dijon Bourgogne, Dijon
  - CHU de Grenoble, La Tronche
  - AP-HP CHU Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHRU,Hôpital Jeanne de Flandres, Lille
  - CHU de Limoges, Limoges
  - AP-HM La Timone, Marseille
  - AP-HM Nord, Marseille
  - CHRU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHR d'Orléans, Orléans
  - AP-HP Armand Trousseau, Paris
  - AP-HP Necker-Enfants malades, Paris
  - AP-HP Robert-Debré, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy
- CHU de Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lejeune S, Sfeir R, Rousseau V, Bonnard A, Gelas T, Aumar M, Panait N, Rabattu PY, Irtan S, Fouquet V, Le Mandat A, Cocci SN, Habonimana E, Lamireau T, Lemelle JL, Elbaz F, Talon I, Boudaoud N, Allal H, Buisson P, Petit T, Sapin E, Lardy H, Schmitt F, Levard G, Scalabre A, Michel JL, Jaby O, Pelatan C, De Vries P, Borderon C, Fourcade L, Breaud J, Arnould M, Tolg C, Chaussy Y, Geiss S, Laplace C, Drumez E, El Mourad S, Thumerelle C, Gottrand F. Esophageal Atresia and Respiratory Morbidity. Pediatrics. 2021 Sep;148(3):e2020049778. doi: 10.1542/peds.2020-049778. Epub 2021 Aug 19. PMID 34413249
- See also: Related Info — http://cracmo.chru-lille.fr/